CLINICAL TRIAL: NCT03885245
Title: Supplementing L-citrulline to Overweight Late Asthma oNset Phenotypes to Increase Airway L-arginine/ADMA Ratio and Improve Asthma Control
Brief Title: Supplementing L-citrulline to Overweight Late Asthma oNset Phenotypes
Acronym: SANDIA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 19-0219; R01HL146542 (NIH)
Record Dates: First submitted 2019-03-06; First posted 2019-03-21 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Asthma; Obesity
MeSH Terms: conditions — Asthma; Obesity | interventions — Citrulline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- L-citrulline (Experimental): L-citrulline with a dose of 15 g/day will be administered in powder form that is mixed with water and taken orally, continuously and daily for at least 7 weeks. Dispensed at Visits 1 and 1a (if needed). Washout period of at least 5 weeks and then enter crossover phase of an additional 7 weeks. Drug will be dispensed at Visit 4.
  Interventions: Drug: L-ctirulline
- Matching Placebo (Placebo Comparator): Administered in powder form that is mixed with water and taken orally, continuously, and daily for at least 7 weeks. Dispensed at Visits 1 and 1a (if needed). Washout period of at least 5 weeks and then enter crossover phase of an additional 7 weeks. Drug will be dispensed at Visit 4.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: L-ctirulline — 7 weeks of treatment with 15 g/day of orally administered (powder form mixed with water) L-citrulline
  Other Names: L-citrulline
  Arms: L-citrulline
Drug: Matching Placebo — 7 weeks of treatment with orally administered matching placebo (to 15 g/day of L-citrulline)
  Arms: Matching Placebo

SUMMARY:
Patients with obese late onset (after childhood) asthma can have lower FeNO levels, yet be highly symptomatic and poorly responsive to inhaled steroids. This is a common asthma phenotype, particularly among females. This reduction of NO occurs through increased arginase activity and uncoupling of NO synthase (NOS), by accumulation of asymmetric di-methyl arginine (ADMA), which further lowers the L-arginine/ADMA ratio, preferentially promoting reactive oxygen species (ROS) formation and inflammation at the expense of NO. Indeed, in patients with obese late onset asthma, lower L-arginine/ADMA plasma ratios are associated with reduced FeNO, increased bronchial hyperreactivity, and greater asthma morbidity. In our pilot studies, the administration of L-citrulline, as an L-arginine donor, to patients with obese late onset asthma increased the L-arginine/ADMA ratio, FeNO levels, and improved asthma control and lung function. Therefore, the objectives of the protocol are to: a) determine the efficacy of L-citrulline, as an add-on treatment to improve the asthma control and lung function in obese late onset asthmatics; b) leverage the use of asthmatic and control cells to further understand obesity-related changes in epithelial airway NO metabolism, and how these changes relate to bronchoconstriction and lung function, c) determine airway epithelial changes in mitochondrial function and bioenergetics in obese late onset asthmatics and how these are modified by L-citrulline. To do this, 54 obese late onset asthmatics with suboptimal control will be blindly randomized, in a cross over study, comparing 15g/day of L-citrulline vs. placebo, in two 8-week treatment periods with a 6-week washout in between. The co-primary study outcomes are asthma control (ACQ, ACT) and FeNO, and secondary endpoints plasma L-arginine/ADMA, FEV1 and PC20 methacholine. Parallel to this study, a small study of 10 healthy obese controls will receive open label L-citrulline for 7 weeks to establish comparative reference values for the study aims. During the initial treatment phase, 50% of study participants will be randomly allocated to undergo pre and post L-citrulline treatment bronchoscopy to obtain BAL and airway epithelial cells. The research group proposing this study is highly experience in asthma clinical trials, implementation of cross over design studies, and in the use of research bronchoscopies.

ELIGIBILITY:
Inclusion Criteria:

1. Adequate completion of informed consent process
2. Male and female patients
3. Physician diagnosis of asthma
4. Able to perform reproducible spirometry according to ATS criteria
5. Pre-bronchodilator FEV1 >/= 50% of predicted at Visit 0
6. Confirmation of asthma
7. All racial/ethnic backgrounds may participate.
8. BMI >/= 30
9. Regular treatment with ICS or ICS/LABA or LAMA combination medication for at least 1 month; participants can be on biologics.
10. Smoking history </= 10 pack years and no smoking in the last 3 months
11. Age of asthma onset (diagnosis) >/= 12 years
12. FeNO </= 30 ppb
13. ACQ >/= 0.50 or ACT </=19

Exclusion Criteria:

1. Respiratory tract infection within the 4 weeks prior to Visit 1
2. Oral or systemic corticosteroid burst (for any indication) within the 4 weeks prior to Visit 0. (One-time doses, such as intra-articular injections into a shoulder or knee joint, require a 4-week washout prior to Visit 0)
3. Asthma-related ER visit within the previous 4 weeks of Visit 0
4. History of ICU admission/intubation due to asthma in the past 1 year
5. 3 or more asthma exacerbations requiring treatment with systemic corticosteroids for more than three days in the past year consistent with severe asthma
6. Asthma exacerbation requiring systemic corticosteroids within the 4 weeks prior to Visit 0.
7. Chronic renal failure
8. Positive urine cotinine or THC test on the day of the bronchoscopy visit
9. Positive urine (or serum) pregnancy test at Visit 0 or at any time during the study
10. Intolerance or allergy to L-arginine or L-citrulline
11. Concomitant use of PDE5 drugs or oral mononitrates
12. Untreated sleep apnea
13. Participant in an interventional drug study or use of investigative drugs within the past 30 days or plans to enroll in such a trial during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Asthma Control Questionnaire | Through study completion, up to 32 weeks
  to determine L-citrulline efficacy, reduction in questionnaire scores determined by administering the questionnaires before, mid-way, and after during each treatment phase to see if there's a change in scores.
Change in Asthma Control Test | Through study completion, up to 32 weeks
  To determine L-citrulline efficacy, reduction in questionnaires scores determined by administering the questionnaires before, mid-way, and after during each treatment phase to see if there's a change in scores.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Holguin, MD, MPH, Principal Investigator — University of Colorado Denver- Anschutz Medical Campus
Locations (1):
- Duke University (Asthma, Allergy and Airway Center), Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No